CLINICAL TRIAL: NCT02869945
Title: Dopaminergic Denervation and COMT Polymorphism in de Novo Patients With Parkinson's Disease
Brief Title: Compensation Mechanisms in Parkinson's Disease
Acronym: DATACOMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P130939
Record Dates: First submitted 2016-08-04; First posted 2016-08-17 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease
Keywords: de novo untreated Parkinson Disease; genetic; COMT Polymorphism; gene; brain MRI; brain MPET
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- COMT HH (Other): COMT HH gene
  Interventions: Genetic: Identification of COMT HH, COMT HL or COMT LL genes; Other: Brain MRI with resting state scan; Other: Brain MPET
- COMT HL (Other): COMT HL gene
  Interventions: Genetic: Identification of COMT HH, COMT HL or COMT LL genes; Other: Brain MRI with resting state scan; Other: Brain MPET
- COMT LL (Other): COMT LL gene
  Interventions: Genetic: Identification of COMT HH, COMT HL or COMT LL genes; Other: Brain MRI with resting state scan; Other: Brain MPET

INTERVENTIONS:
Genetic: Identification of COMT HH, COMT HL or COMT LL genes — COMT HH, COMT HL or COMT LL genes identification
Other: Brain MRI with resting state scan — MRI scan with resting state study to be performed to assess the compensation mechanisms at the networks level.
Other: Brain MPET — Monophotonic emission tomography with I-123-Ioflupane to assess the level of dopaminergic denervation.

SUMMARY:
Parkinson's disease onset is clinically defined as the appearance of motor symptoms including akinesia, tremor and hypertonia. Several studies have shown that motor symptoms occur when at least 50 % of dopaminergic neurons are lost. However, there are evidence suggesting that the level of dopaminergic denervation is not homogenous at the time of diagnosis.

Some patients have a higher level of dopaminergic loss at disease onset indicating the existence of compensation mechanisms. The aim of this study is to decipher how the metabolism of dopamine is involved in this compensation with a focus on the polymorphism of the COMT gene. This gene is expressed according to two variant: (i) COMT H that encodes a form of the enzyme with a high level of activity and (ii) COMT L that encode a form of the enzyme with a low level of activity. Thus, there are 3 possible genotypes in the population: (i) COMT HH associated with an increased degradation of dopamine, (ii) COMT LL associated with a decreased degradation of dopamine and (iii) COMT HH (intermediary between COMT HH and COMT LL).

The hypothesis is that this polymorphism of the COMT gene may participate to compensation mechanisms in early PD. Patients with COMT HH genotype may have an earlier motor symptoms onset than patients with COMT LL genotype.

To test this hypothesis, we will recruit 51 patients with de novo PD will be recruited (17 patients for each genotype). Given the distribution of COMT polymorphism in the population, a maximum sample of 76 patients will be screened to recruit 17 patients for each genotype.

Clinical evaluation will include MDS-UPDRS, Non Motor Symptoms Scale, segmental symptoms scale, Montreal Cognitive assessment, MMSE, Frontal assessment battery and Parkinson's disease behavioral assessment scale (ECMP). All the patients will have a monophotonic emission tomography with I-123-Ioflupane in order to assess the level of dopaminergic denervation and an MRI scan with resting state study. Cerebrospinal fluid sampling will be optional and will allow direct measurements of dopamine metabolites.

The main outcome measure will be the level of dopaminergic denervation on I-123-Ioflupane scans according to COMT genotype, age, gender and severity of motor symptoms on the MDS-UPDRS part 3.

If this hypothesis is confirmed, this will allow to test the efficacy of COMT inhibitors in order to delay dopaminergic drugs initiation for PD patients.

DETAILED DESCRIPTION:
Parkinson's disease onset is clinically defined as the appearance of motor symptoms including akinesia, tremor and hypertonia. Several studies have shown that motor symptoms occur when at least 50 % of dopaminergic neurons are lost. However, there are evidence suggesting that the level of dopaminergic denervation is not homogenous at the time of diagnosis. Some patients have a higher level of dopaminergic loss at disease onset indicating the existence of compensation mechanisms.

The aim of this study is to decipher how the metabolism of dopamine is involved in this compensation with a focus on the polymorphism of the COMT gene. This gene is expressed according to two variants: (i) COMT H that encodes a form of the enzyme with a high level of aactivity and (ii) COMT L that encode a form of the enzyme with a low level of activity. Thus, there are 3 possible genotypes in the population: (i) COMT HH associated with an increased degradation of dopamine, (ii) COMT LL associated with a decreased degradation of dopamine and (iii) COMT HH (intermediary between COMT HH and COMT LL).

The hypothesis is that this polymorphism of the COMT gene may participate to compensation mechanisms in early PD. Patients with COMT HH genotype may have an earlier motor symptoms onset than patients with COMT LL genotype.

To test this hypothesis, 51 patients with de novo PD will be included (17 patients for each genotype). Given the distribution of COMT polymorphism in the population, a maximum sample of 76 patients will be screened for inclusion of 17 patients for each genotype.

Only untreated patients will be included in the study in order to have a reliable assessment of motor severity without interference of dopaminergic drugs.

The study will be scheduled as follow:

* At the first visit (V1), inclusion criteria will be checked and patients will sign the informed consent. COMT genotype of selected patients will be analyzed.
* Result of COMT genotype will be obtained within 4 weeks. Only the 17 first patients with each genotype will continue the study
* For these patients, an evaluation visit with clinical assessment including MDS-UPDRS, Non Motor Symptoms Scale, segmental symptoms scale, Montreal Cognitive assessment, MMSE, Frontal assessment battery and Parkinson's disease behavioral assessment scale (ECMP) will be performed..

All the patients will have a monophotonic emission tomography with I-123-Ioflupane in order to assess the level of dopaminergic denervation. An MRI scan with resting state study will also be performed to assess the compensation mechanisms at the networks level. Cerebrospinal fluid sampling will be optional and will allow direct measurements of dopamine metabolites.

The main outcome measure will be the level of dopaminergic denervation on I-123-Ioflupane scans according to COMT genotype with and without adjustment for age, gender and severity of motor symptoms on the MDS-UPDRS part 3.

Secondary outcome measures will include:

* level of dopaminergic denervation compared across the 3 genotypes (COMT HH, COMT HL and COMT HH) with and without adjustment for age, gender and motor scores
* determination of functional compensation at the networks scale assessed on fMRI resting state scan according to dopaminergic denervation
* determination of CSF dopamine metabolite profile at the time of diagnosis (CSF sampling will be optional).

If this hypothesis is confirmed, this will allow to test the efficacy of COMT inhibitors in order to delay dopaminergic drugs initiation for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years old,
* Caucasian origin
* Parkinson's disease considered to be probable as defined by the criteria of UK Parkinson's disease Brain Bank (Hugues and coll 2002)
* Absence of anti-parkinsonian medication
* Patient affilied to a social security system
* Signed information consent form

Exclusion Criteria:

* Parkinsonian syndrome secondary to neuroleptics
* Atypical parkinsonian syndrome such a multisystem atrophy, progressive supranuclear paralysis, dementia with levy bodies.
* MRI contraindication (claustrophobia, not compatible mechanical heart valve MRI, pacemaker, cochlear implant, other body ferromagnetic objects, pregnancy) - MPET contraindication (pregnancy, feeding, hypersensitivity to ioflupane [123]
* Patient under guardianship or trusteeship
* Any other significant pathology that could prevent patient participation and achievement of planned examinations (except for lumbar puncture)
* Patient participating or having participated in other biomedical research involving a drug in the three months prior to inclusion
* Specific exclusion criteria if lumbar puncture is accepted by the patient: Anticoagulation or antiplatelet treatment; history of hemostasis disorders; platelets <150,000 mm3; TP <80%; TCA (patient / control)> 1.2.
* Hypersensitivity to local anesthetics with amide link or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the degree of presynaptic dopaminergic denervation across the 3 genotypes group (COMT HH, COMT HL and COMT LL) at the time of diagnostic of Parkinson disease | Within 3 months after inclusion
  The degree of presynaptic dopaminergic denervation estimated by the potential links of 123I-FP-CIT (radioligand dopamine transporter) on scintigraphy images of single photon emission

SECONDARY OUTCOMES:
Degree of presynaptic denervation in three groups: COMT HH, COMT LL, COMT HL with and without adjustment for age, sex and UPDRS III score | Within 3 months after inclusion
CSF dopamine metabolite levels at the time of diagnosis (CSF sampling will be optional) in the groups COMT HH, COMT HL and COMT LL | Within 3 months after inclusion
Functional connectivity resting MRI Index obtained by full integration and graph theory based on genotypes (COMT HH, COMT LL, COMT HL) and denervation degree (MPET). | Within 3 months after inclusion
MDS UPDRS-III motor score according to the genotypes (COMT HH, COMT LL, COMT HL) and denervation degree observed by MPET | Within 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: David Grabli, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No